CLINICAL TRIAL: NCT01504308
Title: Philips Pivotal Clinical Trial for MRI-guided High Intensity Focused Ultrasound Ablation of Uterine Fibroids
Brief Title: Sonalleve Fibroid Ablation Pivotal Clinical Trial for MR-HIFU of Uterine Fibroids
Acronym: SOFIA
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: It was not possible to enroll patients into the study in a realistic timeframe.
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 994045; G110008 (Other: FDA)
Record Dates: First submitted 2012-01-03; First posted 2012-01-05 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Uterine Fibroids
Keywords: uterine fibroids; uterine leiomyomas; magnetic resonance imaging; focused ultrasound
MeSH Terms: conditions — Leiomyoma; Myofibroma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- MR-HIFU treatment (Experimental): Patients receiving MR-HIFU treatment
  Interventions: Device: MR-HIFU treatment
- Sham Treatment (Sham Comparator): Patients receiving sham treatment
  Interventions: Device: Sham treatment

INTERVENTIONS:
Device: MR-HIFU treatment — A treatment session with the Philips Sonalleve MR-HIFU device for thermal ablation of uterine fibroids with high-intensity focused ultrasound.
  Other Names: Philips Sonalleve MR-HIFU Uterine Fibroid Therapy
  Arms: MR-HIFU treatment
Device: Sham treatment — A pretend treatment session with the Philips Sonalleve MR-HIFU system in which no therapeutic ultrasound doses are delivered.
  Other Names: pretend treatment with Philips Sonalleve MR-HIFU
  Arms: Sham Treatment

SUMMARY:
The purpose of this clinical study is to determine whether treatment with the Philips Sonalleve Magnetic Resonance-guided High Intensity Focused Ultrasound (MR-HIFU) system is effective in the treatment symptomatic uterine leiomyomas (uterine fibroids).

DETAILED DESCRIPTION:
Uterine Fibroids are the most common benign tumors in pre- and peri-menopausal women. Fibroids occur in 20-50% of women over 30 years of age, and with increasing size can produce pain, menorrhagia, pressure, bloating and urinary and bowel compression symptoms. Fibroids may also cause infertility. Symptomatic fibroids impact health and well-being of the female including lost work hours and reduced quality of life.

Current medical treatments include invasive removal of the fibroid (hysterectomy, myomectomy), drug therapy, or treatments causing necrosis of the fibroid tissue such as ablation (freezing or heating) or embolization. It has been estimated that 600,000 hysterectomies are performed per year in the United States and more than half of the conducted hysterectomies are due to fibroids. For the relief of symptoms, women wishing to preserve the uterus may choose between invasive procedures of myomectomy, Uterine Artery Embolization (UAE), ablation or cryotherapy. The surgically invasive procedures require anesthesia, hospital stays, and long recovery periods. However, High Intensity Focused Ultrasound (HIFU) shows promising results in relieving fibroid symptoms.

This study will confirm the safety and clinical effectiveness of Philips Sonalleve MR-HIFU Fibroid Therapy system for ablating symptomatic fibroids.

ELIGIBILITY:
Inclusion Criteria:

* Women, age between 18 and 50 years
* Ethnicity has a match with the intended profile for the site
* Weight < 140kg or 310lbs
* Pre- or peri-menopausal as indicated by clinical evaluation or Follicle Stimulating Hormone (FSH) level < 40 IU/L
* Willing and able to attend all study visits
* Willing and able to complete Menstrual Blood Loss (MBL) assessment with Alkaline Hematin (AH) method
* Willing and able to use reliable contraception methods
* Uterine size < 24 weeks
* Cervical cell assessment by Pap smear: Normal, Low Grade Squamous Intraepithelial Lesion (SIL), Low risk Human Papillomavirus (HPV) or Atypical Squamous Cells of Uncertain Significance (ASCUS) subtypes of cervical tissue
* MR-HIFU device accessibility to fibroids such that at least 50% of the total fibroid volume can be treated.
* Fibroids selected for treatment meeting the following criteria (further extrapolated in the protocol):

  1. Total planned ablation volume of all fibroids should not exceed 250 ml and
  2. No more than 5 fibroids should be planned for ablation and
  3. Dominant fibroid (diameter) is greater than or equal to 3 cm and
  4. Completely non-enhancing fibroids should not be treated as the identification of treated volume becomes ambiguous
* Patient's self-assessment indicates that she has had episodes of heavy menstrual bleeding in the past 6 months.
* Menstrual Blood Loss (MBL) ≥150 ml and ≤ 500 ml

Exclusion Criteria:

* Other Pelvic Disease (Other mass, endometriosis, ovarian tumor, acute pelvic disease, significant adenomyosis)
* Desire for future pregnancy
* Significant systemic disease even if controlled
* Positive pregnancy test
* Hematocrit < 25%
* Extensive scarring along anterior lower abdominal wall (>50% of area)
* Surgical clips in the potential path of the HIFU beam
* MRI contraindicated
* MRI contrast agent contraindicated (including renal insufficiency)
* Calcifications around or throughout uterine tissues that may affect treatment
* Communication barrier
* Highly perfused or brighter than myometrium in T2-weighted MRI (according to the T2 contrast obtained using the Philips MR-HIFU MR protocol) fibroids
* Fibroids not quantifiable on MRI (e.g. multi-fibroid cases where volume measurements are not feasible)
* Menses lasting > 7 days or intermenstrual bleeding (patient can be included if there is endometrial biopsy within 6 months to exclude malignancy)
* Patient is currently on hormonal medication for fibroids or has a hormonal medication history as described below:

  1. 1-month Lupron dose or equivalent: less than 1 month prior to MBL measurement or
  2. 3-month Lupron dose or equivalent: less than 3 months prior to MBL measurement or
  3. Depo Provera or equivalent: less than 6 months prior to MBL measurement

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2012-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Alternative Interventional Treatment (AIT) | 12 months after HIFU treatment
  AIT is scored dichotomously as follows:
  0 = Failure. Failure occurs if an AIT for fibroid related symptoms is administered within 12 months of study treatment.
  1 = Success. Success occurs if no AIT is administered for fibroid related symptoms within 12 months of study treatment.
  An AIT is defined as being one of the following: hysterectomy, myomectomy, uterine artery embolization, endometrial ablation and resection, or another MR-HIFU treatment (with the exception of a 're-treatment' as defined in the protocol, e.g. because of temporarily inaccessible fibroids).
Menstrual Blood Loss (MBL) | at baseline and at 12 months following treatment
  Menstrual Blood Loss (MBL) scored dichotomously as follows:
  0 = Failure. Failure occurs if the change from baseline in MBL measurement is < 50 % as measured with alkaline hematin test (AHT) method.
  1 = Success. Success occurs if the change from baseline in MBL measurement is >= 50 %, or if the MBL is < 80 ml as measured with the AHT method.

SECONDARY OUTCOMES:
Return to Activity | 72 hours
  Length for Return to Activity after HIFU treatment measured dichotomously:
  0 = Failure. If subject takes longer than 72 hours to return to work or normal activity.
  1 = Success. If subject returns to work or normal activity within 72 hours inclusive.
Symptom Severity Score (SSS) | at baseline and at 12 months following treatment
  Symptom Severity Score (SSS) of Uterine Fibroid Symptom and Quality of Life questionnaire (UFS-QoL), assessed dichotomously at 12 months:
  0 = Failure. Reduction of less than 10 points on SSS.
  1 = Success. Reduction of at least 10 points on SSS.

CONTACTS AND LOCATIONS:
Overall Officials: John H Fischer II, MD, Principal Investigator — St. Luke's Episcopal Hospital, Houston, Texas, United States; Robert K Zurawin, MD, Principal Investigator — St. Luke's Episcopal Hospital, Houston, Texas, United States; Elizabeth David, MD, Principal Investigator — Sunnybrook Health Sciences Center, Toronto, Ontario, Canada; Hyo Keun Lim, MD, Principal Investigator — Samsung Medical Center, Seoul, Republic of Korea; Aytekin Oto, MD, Principal Investigator — University of Chicago, Chicago, Illinois, United States; Amanda Yunker, D.O., Principal Investigator — Vanderbilt Medical Center; Peter Liu, M.D., Principal Investigator — University of Michigan; Rajiv Chopra, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (9):
- United States (7):
  - University of Chicago, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Montefiore Medical Center, The Bronx, New York
  - Oregon Science and Health University, Portland, Oregon
  - Vanderbilt Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Voogt MJ, Trillaud H, Kim YS, Mali WP, Barkhausen J, Bartels LW, Deckers R, Frulio N, Rhim H, Lim HK, Eckey T, Nieminen HJ, Mougenot C, Keserci B, Soini J, Vaara T, Kohler MO, Sokka S, van den Bosch MA. Volumetric feedback ablation of uterine fibroids using magnetic resonance-guided high intensity focused ultrasound therapy. Eur Radiol. 2012 Feb;22(2):411-7. doi: 10.1007/s00330-011-2262-8. Epub 2011 Sep 8. PMID 21901565
- [Background] Spies JB, Coyne K, Guaou Guaou N, Boyle D, Skyrnarz-Murphy K, Gonzalves SM. The UFS-QOL, a new disease-specific symptom and health-related quality of life questionnaire for leiomyomata. Obstet Gynecol. 2002 Feb;99(2):290-300. doi: 10.1016/s0029-7844(01)01702-1. PMID 11814511
- [Background] Stewart EA, Gedroyc WM, Tempany CM, Quade BJ, Inbar Y, Ehrenstein T, Shushan A, Hindley JT, Goldin RD, David M, Sklair M, Rabinovici J. Focused ultrasound treatment of uterine fibroid tumors: safety and feasibility of a noninvasive thermoablative technique. Am J Obstet Gynecol. 2003 Jul;189(1):48-54. doi: 10.1067/mob.2003.345. PMID 12861137
- [Background] Hindley J, Gedroyc WM, Regan L, Stewart E, Tempany C, Hynyen K, Mcdannold N, Inbar Y, Itzchak Y, Rabinovici J, Kim HS, Geschwind JF, Hesley G, Gostout B, Ehrenstein T, Hengst S, Sklair-Levy M, Shushan A, Jolesz F. MRI guidance of focused ultrasound therapy of uterine fibroids: early results. AJR Am J Roentgenol. 2004 Dec;183(6):1713-9. doi: 10.2214/ajr.183.6.01831713. PMID 15547216
- [Background] Leon-Villapalos J, Kaniorou-Larai M, Dziewulski P. Full thickness abdominal burn following magnetic resonance guided focused ultrasound therapy. Burns. 2005 Dec;31(8):1054-5. doi: 10.1016/j.burns.2005.04.019. Epub 2005 Jun 20. No abstract available. PMID 15970389
- [Background] Fennessy FM, Tempany CM. MRI-guided focused ultrasound surgery of uterine leiomyomas. Acad Radiol. 2005 Sep;12(9):1158-66. doi: 10.1016/j.acra.2005.05.018. PMID 16099686
- [Background] Stewart EA, Rabinovici J, Tempany CM, Inbar Y, Regan L, Gostout B, Hesley G, Kim HS, Hengst S, Gedroyc WM. Clinical outcomes of focused ultrasound surgery for the treatment of uterine fibroids. Fertil Steril. 2006 Jan;85(1):22-9. doi: 10.1016/j.fertnstert.2005.04.072. PMID 16412721
- [Background] Fennessy FM, Tempany CM, McDannold NJ, So MJ, Hesley G, Gostout B, Kim HS, Holland GA, Sarti DA, Hynynen K, Jolesz FA, Stewart EA. Uterine leiomyomas: MR imaging-guided focused ultrasound surgery--results of different treatment protocols. Radiology. 2007 Jun;243(3):885-93. doi: 10.1148/radiol.2433060267. Epub 2007 Apr 19. PMID 17446521
- [Background] Mara M, Fucikova Z, Maskova J, Kuzel D, Haakova L. Uterine fibroid embolization versus myomectomy in women wishing to preserve fertility: preliminary results of a randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2006 Jun 1;126(2):226-33. doi: 10.1016/j.ejogrb.2005.10.008. Epub 2005 Nov 15. PMID 16293363
- [Background] Stewart EA, Gostout B, Rabinovici J, Kim HS, Regan L, Tempany CM. Sustained relief of leiomyoma symptoms by using focused ultrasound surgery. Obstet Gynecol. 2007 Aug;110(2 Pt 1):279-87. doi: 10.1097/01.AOG.0000275283.39475.f6. PMID 17666601
- [Background] Taran FA, Tempany CM, Regan L, Inbar Y, Revel A, Stewart EA; MRgFUS Group. Magnetic resonance-guided focused ultrasound (MRgFUS) compared with abdominal hysterectomy for treatment of uterine leiomyomas. Ultrasound Obstet Gynecol. 2009 Nov;34(5):572-8. doi: 10.1002/uog.7435. PMID 19852046
- [Background] Funaki K, Fukunishi H, Sawada K. Clinical outcomes of magnetic resonance-guided focused ultrasound surgery for uterine myomas: 24-month follow-up. Ultrasound Obstet Gynecol. 2009 Nov;34(5):584-9. doi: 10.1002/uog.7455. PMID 19852041
- [Background] Okada A, Morita Y, Fukunishi H, Takeichi K, Murakami T. Non-invasive magnetic resonance-guided focused ultrasound treatment of uterine fibroids in a large Japanese population: impact of the learning curve on patient outcome. Ultrasound Obstet Gynecol. 2009 Nov;34(5):579-83. doi: 10.1002/uog.7454. PMID 19852042
- [Background] Kim YS, Lim HK, Kim JH, Rhim H, Park BK, Keserci B, Kohler MO, Bae DS, Kim BG, Lee JW, Kim TJ, Sokka S, Lee JH. Dynamic contrast-enhanced magnetic resonance imaging predicts immediate therapeutic response of magnetic resonance-guided high-intensity focused ultrasound ablation of symptomatic uterine fibroids. Invest Radiol. 2011 Oct;46(10):639-47. doi: 10.1097/RLI.0b013e318220785c. PMID 21654495